CLINICAL TRIAL: NCT02883335
Title: Lorraine Registry of Multiple Sclerosis
Acronym: RelSEP
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Lorraine (Other)
Responsible Party: Principal Investigator, GUILLEMIN Francis, MD, Médecine coordonateur de module, Central Hospital, Nancy, France
Other Study IDs: RELSEP
Record Dates: First submitted 2016-08-19; First posted 2016-08-30 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Observational registry

SUMMARY:
The RelSEP aims to register exhaustively every new case of multiple sclerosis (MS) occuring in Lorraine a French region, and follow up on them for an indefinite duration, registering disease evolution and intercurrent events.

DETAILED DESCRIPTION:
As every patient registry in France, the RelSEP is periodically (every four years) evaluated by an independent committee.

The RelSEP interrogate multiple sources to insure its exhaustiveness :

* every neurologists of Lorraine
* MS patient network in Lorraine
* health insurance data
* PMSI (administrative French national database for hospitals)
* biological and imagery services in Lorraine Procedures (automatic and manual) are used to eliminate duplicates Once a patient has been identified its medical file are checked by investigators in order to retrieve the relevant information.

New MS cases are confirmed by neurologists. Automatics (implemented in EDMUS software)and manual checks are implemented in the registry database, looking for inconsistencies.

The following data are registered :

* Name, birthname
* Sex
* Date of birth
* Location (town)
* Birth location (town)
* Profession
* Number of siblings
* Marital status
* Number of children
* Date of onset
* Date and nature of clinical manifestations
* MRI reports
* CSF analysis reports
* Event-related potential reports
* Impairment and disability evolution
* Treatments (start and change of drug treatment)
* Drugs related events
* Cause of treatment discontinuation
* Disease progression Every case has a follow up at least every two years.

The quality of data is evaluated by periodically auditing cases at random from our database.

An annual report on the main data (incidence and prevalence) of MS in Lorraine is produced.

Data are also used for observational studies on prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* Having a confirmed multiple sclerosis diagnosis
* Living in Lorraine (French region)

Exclusion Criteria:

* Refusal to be registered

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from multiple sclerosis in Lorraine
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2003-05; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
case occurence of multiple sclerosis | one year

SECONDARY OUTCOMES:
EDSS score | 30 years

CONTACTS AND LOCATIONS:
Overall Officials: Francis Guillemin, MD, PHD, Principal Investigator — CHRU Nancy
Locations (1):
- CIC 1433 Épidémiologie clinique, Inserm, Université de Lorraine, CHRU de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: Yes
open to partnership

REFERENCES:
- [Background] Brissart H, Morele E, Baumann C, Perf ML, Leininger M, Taillemite L, Dillier C, Pittion S, Spitz E, Debouverie M. Cognitive impairment among different clinical courses of multiple sclerosis. Neurol Res. 2013 Oct;35(8):867-72. doi: 10.1179/1743132813Y.0000000232. Epub 2013 Jun 19. PMID 23816638
- [Background] Brissart H, Sauvee M, Latarche C, Dillier C, Debouverie M. Integration of cognitive impairment in the expanded disability status scale of 215 patients with multiple sclerosis. Eur Neurol. 2010;64(6):345-50. doi: 10.1159/000322140. Epub 2010 Nov 13. PMID 21071951
- [Result] El Adssi H, Debouverie M, Guillemin F; LORSEP Group. Estimating the prevalence and incidence of multiple sclerosis in the Lorraine region, France, by the capture-recapture method. Mult Scler. 2012 Sep;18(9):1244-50. doi: 10.1177/1352458512437811. Epub 2012 Feb 21. PMID 22354740
- [Result] Becker M, Latarche C, Roman E, Debouverie M, Malaplate-Armand C, Guillemin F. No prognostic value of routine cerebrospinal fluid biomarkers in a population-based cohort of 407 multiple sclerosis patients. BMC Neurol. 2015 May 13;15:79. doi: 10.1186/s12883-015-0330-4. PMID 25966681